CLINICAL TRIAL: NCT04215614
Title: The Comparison of Lateral Sagittal vs Costoclavicular Brachial Plexus Block in Children
Brief Title: Lateral Sagittal vs Costoclavicular Brachial Plexus Block in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LS vs Costo BPB Pediatric
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hand Injuries and Disorders; Forearm Injuries
MeSH Terms: conditions — Hand Injuries; Disease; Forearm Injuries | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lateral Sagittal (Active Comparator): Ultrasound-Guided lateral sagittal brachial plexus block with 1:1 ratio 2% lidocaine, and 0.5% bupivacaine
  Interventions: Drug: Lidocaine and Bupivacaine solution; Device: Lateral Sagittal block
- Group Costoclavicular (Active Comparator): Ultrasound-Guided costoclavicular brachial plexus block with 1:1 ratio 2% lidocaine, and 0.5% bupivacaine
  Interventions: Drug: Lidocaine and Bupivacaine solution; Device: Costoclavicular block

INTERVENTIONS:
Drug: Lidocaine and Bupivacaine solution — 1:1 ratio 2% lidocaine, and 0.5% bupivacaine
Device: Costoclavicular block — Ultrasound-guided costoclavicular brachial plexus block
  Arms: Group Costoclavicular
Device: Lateral Sagittal block — Ultrasound-guided lateral sagittal brachial plexus block
  Arms: Group Lateral Sagittal

SUMMARY:
Costoclavicular approach has lots of advantages compared to the lateral sagittal approach for infraclavicular brachial plexus block. Although the efficacy of this block has been demonstrated in adults, there are no randomized controlled trials in the literature on the application of pediatric patients. Our aim was to compare the ultrasound-guided infraclavicular and costoclavicular approach in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients
* Patients who will undergo hand or forearm surgery

Exclusion Criteria:

* Infection in the area to be injected
* Coagulopathy,
* Previously known neurological damage

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Block performance time | Twenty minutes before surgery
  The time interval between the contact of the ultrasound probe to skin and end of local anesthetics injection.

SECONDARY OUTCOMES:
Visual analog pain score | Postoperative 24 hours
  Pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Yayik AM, Cesur S, Ozturk F, Celik EC, Ahiskalioglu A. Ultrasound guided costoclavicular approach to brachial plexus: First pediatric report. J Clin Anesth. 2019 Aug;55:136-137. doi: 10.1016/j.jclinane.2019.01.008. Epub 2019 Jan 15. No abstract available. PMID 30658327
- [Background] Songthamwat B, Karmakar MK, Li JW, Samy W, Mok LYH. Ultrasound-Guided Infraclavicular Brachial Plexus Block: Prospective Randomized Comparison of the Lateral Sagittal and Costoclavicular Approach. Reg Anesth Pain Med. 2018 Nov;43(8):825-831. doi: 10.1097/AAP.0000000000000822. PMID 29923950